CLINICAL TRIAL: NCT02803905
Title: A Monocentric, Open-label, Double-arm, Phase II Trial to Assess the Safety and Efficacy of Allogeneic Islet Cells Transplanted Into the Omentum
Brief Title: Islet Transplant Alone in OMENtum
Acronym: ITA-OMEN
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lorenzo Piemonti (Other)
Responsible Party: Sponsor-Investigator, Lorenzo Piemonti, Deputy director San Raffaele Diabetes Research Institute (SR-DRI), Ospedale San Raffaele
Organization: Ospedale San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITA OMEN
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Islets of Langerhans Transplantation; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- standard procedure: intrahepatic (Active Comparator): Liver infusion: the islet mixture is delivered slowly via injection through a syringe attached to the catheter in the portal vein or portal vein tributary. Access to the portal vein is achieved by percutaneous transhepatic access under fluoroscopic, ultrasonographic, or real-time CT guidance. Alternatively access to a mesenteric or omental venous tributary of the portal vein can be obtained by mini-laparotomy under general anesthesia (transplant site preference or in the extremely rare circumstance that percutaneous access cannot be achieved). At a minimum, portal pressure will be monitored before and after infusion of the islet product. Portal pressure measurements will be documented in the medical record. Gel foam plugs and/or collagen/thrombin paste will be used to embolize the entire peripheral catheter tract immediately before the catheter is withdrawn, to reduce the chances of bleeding.
  Interventions: Biological: Biological: Islet transplantation
- experimental procedure: omentum (Experimental): Omentum infusion: briefly, islets are spread in the surface of the omentum, in a single omental pouch site. Transplanting in a single site will reduce risks. A single dose of at least 5000 IEQ/KG will be transplanted. The investigators should be able to achieve a meaningful metabolic improvement and prevention of severe hypoglycemia, as previously seen in experience with intraportal islet transplants. Recombinant human thrombin is added to the islets placed on the omentum to promote formation of a gel clot and facilitate adherence to the surface of the omentum. A pouch is then created by folding the omentum. The pouch is secured inn place with stitches.
  Interventions: Biological: Biological: Islet transplantation

INTERVENTIONS:
Biological: Biological: Islet transplantation — This is a single procedure protocol. Only a single islet transplant will be performed in the patient. Islets can be isolated from more than one pancreas donor. The final islet product is a sterile suspension of ≥70% viable, ≥30% pure, allogeneic islets. A minimum of 5000 IEQ/KG will be transplanted. Although this study is a single dose protocol, islet transplant recipients with partial islet graft function will be considered for a second islet transplant (intra-hepatic administration) if they do not achieve primary efficacy endpoint criteria at 1 year

SUMMARY:
The study is a phase 2, monocentric, open-label study. The investigators will recruit 12 patients with T1D to be randomly (1:1) assigned to receive islet either into the liver through the portal venous circulation (standard procedure; arm A, n=6) or directly into the omentum (arm B, n=6). Patients will be selected from those eligible for islet Tx based on local practice and guidelines. Immunosuppression will consist of five doses IV infusion of rabbit Anti-thymocyte Globulin (ATG, Thymoglobulin®), starting two days prior to the islet transplant. Maintenance mycophenolate mofetil (MMF) therapy (1-2 g/day as BID dosing) will be started on Day -1 pre-transplant. Tacrolimus will be administered orally twice daily on Day 1 post-transplant to maintain a trough level of 10-12 ng/mL for 3 months, then 6-10 ng/mL thereafter. Etanercept will be given IV before the islet transplant (50 mg), and then at 25 mg (subcutaneously) on POD +3, +7 and +10.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with T1D with onset of disease at <40 years of age, insulin-dependence for > 5 years at the time of enrollment, and a sum of subject age and insulin-dependent diabetes duration of ≥28.
* Absent stimulated c-peptide (<0.3ng/mL) in response to a MMTT
* Involvement in intensive diabetes management
* At least one episode of severe hypoglycemia in the 12 months prior to study enrollment.
* Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more OR a HYPO score greater than or equal to the 90th percentile (1047) during the screening period; OR marked glycemic lability characterized by wide swings in BG despite optimal diabetes therapy and defined by an LI score greater than or equal to the 90th percentile (43 mmol/L2/h·wk-1) during the screening period; OR a composite of a Clarke score of 3 or less and a HYPO score greater than or equal to the 75th percentile (423) and a LI greater than or equal to the 75th percentile (329) during the screening period.

Exclusion Criteria:

* Body Mass Index (BMI) >30 kg/m2 or patient weight ≤50 kg.
* Insulin requirement of >1.0 IU/kg/day or <15 U/day.
* HbA1c >10%.
* Untreated proliferative diabetic retinopathy.
* Blood Pressure: SBP >160 mmHg or DBP >100 mmHg.
* Measured glomerular filtration rate <80 mL/min/1.73 m2.
* Presence or history of macroalbuminuria (>300mg/g creatinine).
* Presence or history of panel-reactive anti-HLA antibodies above background by flow cytometry.
* For female subjects: Serum or urine Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation.
* For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception.
* Presence or history of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
* Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
* Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection within one year prior to study enrollment.
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
* Baseline Hb below the lower limits of normal at the local laboratory; lymphopenia (<1,000/µL), neutropenia (<1,500/µL), or thrombocytopenia (platelets <100,000/µL)
* A history of Factor V deficiency.
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after transplantation (low-dose aspirin treatment is allowed) or patients with an international normalized ratio (INR) >1.5.
* Severe co-existing cardiac disease
* Persistent elevation of liver function tests at the time of study entry.
* Symptomatic cholecystolithiasis.
* Acute or chronic pancreatitis.
* Symptomatic peptic ulcer disease.
* Hyperlipidemia despite medical therapy
* Receiving treatment for a medical condition requiring chronic use of systemic steroids, except for the use of ≤5 mg prednisone daily, or an equivalent dose of hydrocortisone, for physiological replacement only.
* Treatment with any anti-diabetic medications other than insulin within 4 weeks of enrollment.
* Use of any investigational agents within 4 weeks of enrollment. 24. Administration of live attenuated vaccine(s) within 2 months of enrollment.
* Inflammatory bowel disease.
* History of intestinal obstructions.
* Previous major abdominal surgery.
* History of peritonitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
A1c </= 6.5% and no severe hypoglycemia | 1 year
  composite outcome: Proportion of subjects with HbA1c ≤6.5% at 1 year AND free of severe hypoglycemic events from Day 28 to Day 365, inclusive, after the islet transplant.

SECONDARY OUTCOMES:
Insulin requirements | At 75±7, 365 ± 14 ,and 730 ± 14 days following the islet transplant
  the percent reduction in insulin requirements
Insulin secretion | At 75±7, 365 ± 14 ,and 730 ± 14 days following the islet transplant
  basal (fasting) and 90-min glucose and c-peptide derived from the mixed-meal tolerance test (MMTT)
Glucose control | At 75±7, 365 ± 14 ,and 730 ± 14 days following the islet transplant
  HbA1c
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 1 year
  incidence of post-transplant infections, malignancies, morbidity, and other AEs

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Piemonti, MD, Principal Investigator — Ospedale San Raffaele
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Italy